CLINICAL TRIAL: NCT04814329
Title: Study on Predicting Response of Recurrent Glioblastoma to Apatinib
Brief Title: Glioblastoma Response Prediction to Apatinib
Status: Completed | Type: Observational
Sponsor: Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Junping Zhang, Chief physician, Beijing Sanbo Brain Hospital
Other Study IDs: 2021ZZLX03
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Glioblastoma
Keywords: Vascular Endothelial Growth Factor Receptor 2; Biomarkers; glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- effective group: After treatment, tumor achieved complete response or partial response and the progression-free survival time was ≥6 months.
  Interventions: Other: genetic characteristic
- stable group: After treatment, tumor remains stable and the progression-free survival time was more than 1 month and less than 6 months.
  Interventions: Other: genetic characteristic
- Early progressed group: After treatment, tumor got progressed and the progression-free survival time was no more than 1 month.
  Interventions: Other: genetic characteristic

INTERVENTIONS:
Other: genetic characteristic — the underlying genetic characteristics that prodicting response

SUMMARY:
Anti-angiogenic therapy is an important treatment strategy for recurrent glioblastoma. Our previous study provided evidence for a potential benefit of apatinib, a humanized monoclonal antibody against VEGFR-2, when added to temozolomide chemotherapy in patients with recurrent glioblastoma. Some patients showed durable responses and prolonged survival, with recorded survival times of over 30 months in 6.4% patients. However, a subset of patients progressed in 2 months. There is a strong need to better predict and monitor apatinib treatment response to prevent patients from adverse effects of ineffective therapy. In this study, whole genome sequencing and RNA-sequencing of formalin-fixed, paraffin-embedded tumor materials from the participants who received apatinib and temozolomide treatment will be performed to identify the response biomarkers and patients who may benefit most from apatinib, avoiding unnecessary potential toxicity and cost for those who are unlikely to benefit from the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old
2. recurrent glioblastoma
3. received apatinib plus temozolomide treatment，response and survival data were available
4. tumor tissues were acquired

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neuro-oncology Department, Sanbo Bran Hospital Capital Medical University
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
genetic outcome | up to 2 years
  response prodicting biomarker

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University Sanbo Brain Hospital, Beijing, China